CLINICAL TRIAL: NCT03780179
Title: Measles-mumps-rubella Vaccine at 6 Months of Age, Immunology, and Childhood Morbidity in a High-income Setting
Brief Title: MMR at 6 Months Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Lone Graff Stensballe, Pediatrician, associate professor, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LGS.MMR.01.2016.2022
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Meales-mumps-rubella Vaccine
Keywords: measles-mumps-rubella vaccine

STUDY DESIGN:
Intervention Model Description: Randomization to intervention: MMRvaxpro at 6 months of age, or placebo-vaccine (solvent only)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MMRvaxpro (Experimental)
  Interventions: Biological: MMRvaxpro
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MMRvaxpro — MMRvaxpro vaccine
  Arms: MMRvaxpro
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Randomised, double-blind clinical trial to test humoral and cellular immunogenicity, and potential in-direct beneficial effect of the MMRvaxpro-vaccine administered at 6 months of age

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of 32+ weeks.
* Birth weight of 1000+ grams.
* Signed informed consent from the parents.

Exclusion Criteria:

* Immune-deficiency (primary or acquired) or -suppression.
* Intake of immune modulating medicine (including high doses of corticosteroids) (M-M-RVAXPRO is not contraindicated in individuals who are receiving topical or low-dose parenteral corticosteroids, e.g. for asthma prophylaxis or replacement therapy).
* Signs of severe illness or major malformation.
* No Danish-speaking parent.
* Children with a history of anaphylactic, anaphylactoid, or other immediate reactions (e.g., hives, swelling of the mouth and throat, difficulty breathing, hypotension, or shock) subsequent to egg ingestion are excluded.
* Children with known fructose intolerance, thrombocytopenia or any coagulation disorder will be excluded.
* Children who received blood or plasma transfusions, or administration of human immune serum globulin within the last 3 months will be excluded.
* Further, children are excluded from the trial if any contraindication is suspected: history of hypersensitivity to any measles, mumps, or rubella vaccine, or to any of the excipients, including neomycin.
* Children with active untreated tuberculosis, blood dyscrasias, leukaemia, lymphomas of any type, or other malignant neoplasms affecting the haematopoietic and lymphatic systems will be excluded.

Ages: 5 Months to 7 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6540 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Humoral immunogenicity | 1 months after intervention
  The plaque reduction neutralisation test (PRNT), which measures the serum dilution capable of preventing 50% of plaque formation induced by measles virus in cell cultures, has been considered the most reliable criterion for the serologic evaluation of measles immunity. For PNRT, the protective cutoff titer is defined to be >120. A frequency of 95% seroconversion rate, i.e. children mounting a protective level of humoral immunity according to the abovementioned cutoff value after MMR-vaccination at 6 M of age will be considered sufficient to suggest implementation of MMR at 6 M in the Danish vaccination programme.
Hospitalisation for infection | 6-12 months of age
  Significant decrease in hospitalisation for infection measured as repeated events from 6 to 12 months of age in children randomised to MMR at 6 M compared to children randomised to placebo. Information about hospitalisation for infection will be obtained from the national Danish Patient Register, where all Danish inhabitants are followed-up during all hospital contacts.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen, Copenhagen Ø
  - Herlev Hospital, Herlev

REFERENCES:
- [Derived] Buus S, Vittrup DM, Schmidt JD, Jensen A, Stryhn A, Stensballe LG. Measles-mumps-rubella-vaccination at 6 months of age induces measles-specific T cell responses: a randomized controlled trial. Front Immunol. 2025 Mar 17;16:1546253. doi: 10.3389/fimmu.2025.1546253. eCollection 2025. PMID 40165977
- [Derived] Sorensen JK, Jensen A, Zimakoff AC, Vittrup DM, Malon M, Kim S, Hatley EV, Bybjerg-Grauholm J, Kaur S, Pociot F, Stensballe LG, Svensson J. Genetic associations with measles PRNT and IgG antibody response to MMR vaccination in 6- and 15-month-old children. Vaccine. 2025 Mar 19;50:126788. doi: 10.1016/j.vaccine.2025.126788. Epub 2025 Feb 5. PMID 39914254
- [Derived] Vittrup DM, Jensen A, Sorensen JK, Zimakoff AC, Malon M, Charabi S, Johansen MR, Simoes EAF, Kirkby NS, Buus S, Svensson J, Stensballe LG. Immunogenicity and reactogenicity following MMR vaccination in 5-7-month-old infants: a double-blind placebo-controlled randomized clinical trial in 6540 Danish infants. EClinicalMedicine. 2024 Jan 12;68:102421. doi: 10.1016/j.eclinm.2023.102421. eCollection 2024 Feb. PMID 38292039
- [Derived] Zimakoff AC, Jensen A, Vittrup DM, Herlufsen EH, Sorensen JK, Malon M, Svensson J, Stensballe LG. Measles, mumps, and rubella vaccine at age 6 months and hospitalisation for infection before age 12 months: randomised controlled trial. BMJ. 2023 Jun 7;381:e072724. doi: 10.1136/bmj-2022-072724. PMID 37286215